CLINICAL TRIAL: NCT06750848
Title: Chidamide Combined With Angiogenesis Inhibitors and Fulvestrant for Advanced HR-positive, HER2-negative Breast Cancer After Prior CDK4/6 Inhibitor Progression : a Single Arm, Phase Ⅱ Study
Brief Title: Chidamide Combined With Angiogenesis Inhibitors and Fulvestrant for Advanced HR-positive, HER2-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jundong Wu (Other)
Responsible Party: Sponsor-Investigator, Jundong Wu, Affiliated Cancer Hospital of Shantou University Medical College, Affiliated Cancer Hospital of Shantou University Medical College
Organization: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C31
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide，Fulvestrant ，angiogenesis inhibitors (Experimental)
  Interventions: Drug: Chidamide，Fulvestrant，angiogenesis inhibitors

INTERVENTIONS:
Drug: Chidamide，Fulvestrant，angiogenesis inhibitors — chidamide，30mg，po. biw fulvestrant ，500mg， im., d1(c1d15), q4w angiogenesis inhibitors , according to the doctor's advice

SUMMARY:
This Phase Ⅱ study was designed to assess the efficacy and safety of the combination of tucidinostat, angiogenesis inhibitors and fulvestrant for advanced HR-positive, HER2-negative breast cancer patients after the failure of CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age≥18 years, ≤75, female; 2.Histologically confirmed HR positive and HER2 negative postmenopausal metastatic breast cancer patients [HER2 negative is defined as immunohistochemistry(IHC) 0 or IHC 1+, and if the score of IHC is 2+, fluorescence in situ hybridization technology (FISH) test must be negative, HR positve is defined as ER or PR ≥10%]; 3.Prior CDK4/6 inhibitor progression or intolerance to CDK4/6i before enrollment; 4.Premenopausal patients need OFS; 5.Recurrence and metastasis progressed more than 6 months after receiving endocrine therapy or more than 2 years after receiving adjuvant endocrine therapy; 6.ECOG performance status ≤ 1; 7.At least one measurable disease based on RECIST v1.1 8.Adequate organ function; 9.Life expectancy is more than 3 months; 10.Willing and able to provide written informed consent

Exclusion Criteria:

* 1.Prior exposed to histone deacetylase inhibitors; 2.Received TKI before enrollment; 3.Exist visceral crisis; 4.Received chemotherapy, targeted therapy, Chinese herbal medicine with anti-tumor indications, or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 4 weeks before enrollment, or still within 5 half-lives of such drugs; 5.Poorly controlled diabetes (FBG>10mmol/L); 6.Poorly controlled hypertension (SBP>150 mmHg, DBP>90 mmHg); 7.Urinalysis shows urine protein ≥ 2+ or 24-hour protein quantity test shows urinary protein ≥1 g; 8.PT>16s, APTT> 43s, TT>21s, FIB<2g/L; 9.Toxicities that did not recover to National Cancer Institute Common Adverse Event Terminology Version 5.0 (NCICTCAEv5.0) grade 0 or 1 toxicity from prior antineoplastic therapy prior to the first dose of study treatment(alopecia, grade 2 fatigue, grade 2 anemia, non-clinically critical and asymptomatic laboratory abnormalities can be enrolled); 10.Pregnant or lactating female. 11.Any other conditions deemed inappropriate by the investigator to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  Objective Response Rate（ORR）by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Time from treatment until disease progression or death
Disease Control Rate （DCR） | 2 years
  he total proportion of patients with complete response（CR）, partial response（PR）and stable disease（SD）
Clinical Benefit Rate (CBR) | 2 years
  The total proportion of patients with Partial Response (PR), Complete Response (CR) or Stable Disease (SD) ≥6 months
Overall survival (OS) | 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: caiwen du, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center; jundong wu, Principal Investigator — Affiliated Tumor Hospital of Shantou University Medical College
Locations (1):
- Affiliated Tumor Hospital of Shantou University Medical College, Shantou, China

IPD SHARING:
Plan to Share IPD: No